CLINICAL TRIAL: NCT02379806
Title: Prevention of Symptomatic Venous Thromboembolism by Low Molecular Weight Heparin in Hospitalized Medical Patients Aged 70 Years and Older : a Randomized Placebo-Controlled Study The SYMPTOMS (SYstematic Elderly Medical Patients Thromboprophylaxis : Efficacy on Symptomatic OutcoMeS) Study
Brief Title: The SYMPTOMS - SYstematic Elderly Medical Patients Thromboprophylaxis: Efficacy on Symptomatic OutcoMeS - Study
Acronym: SYMPTOMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 29BRC14.0012 SYMPTOMS; 2014-000311-13 (EudraCT Number)
Record Dates: First submitted 2015-02-16; First posted 2015-03-05 (Estimated); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active enoxaparin 40 mg (Active Comparator): One 0.4 ml prefilled syringe containing 40 mg enoxaparin active substance administered once daily for 10 ± 4 days
  Interventions: Drug: Enoxaparin
- Placebo of enoxaparin 40 mg (Placebo Comparator): One 0.4 ml placebo syringe of enoxaparin 40 mg administered once daily for 10 ± 4 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enoxaparin
  Other Names: Lovenox
  Arms: Active enoxaparin 40 mg
Drug: Placebo
  Arms: Placebo of enoxaparin 40 mg

SUMMARY:
Venous thromboembolism (VTE) is a frequent condition, affecting 1.8 per 1,000 people every year. Admission to hospital is one of the main risk factors for VTE, and could account for up to 20% of all VTE, making VTE prevention in admitted patients an appealing option to reduce VTE global burden.

The landmark MEDENOX trial and others demonstrated the efficacy of low molecular weight heparins (LMWH) in reducing a composite outcome of symptomatic and asymptomatic events, the latter accounting for the vast majority of events.

Publication of these trials led to the implementation of thromboprophylaxis policies in hospitals, which acceptance has been variable. More recently, the use of thromboprophylaxis has been challenged after the publication of 1) a negative trial that used 'death from any cause' as main outcome, 2) a systematic review showing the lack of a clear efficacy on the risk of pulmonary embolism or death, 3) negative trials using new oral anticoagulants, 4) the last version of the American College of Chest Physicians Guidelines, focusing on symptomatic events only, downgraded its recommendation for thromboprophylaxis in medical patients to a 1B recommendation, restricting its use to patients 'at increased risk of thrombosis' and recommending against the use of thromboprophylaxis in patients at low risk of thrombosis, patients bleeding or at high risk of bleeding.

However, a limitation of this interpretation of the data is that in most trials, patients with screened asymptomatic events were treated with anticoagulants, preventing the occurrence of symptomatic events during follow-up. Moreover, subgroup analyses showed that elderly patients were at high risk of thrombosis in these trials, and that LMWH could be particularly efficient in this subgroup of patients. Conversely, their risk of bleeding is also higher than in younger patients and the current trials were not powered to detect a difference in the bleeding risk between groups. Finally, the diagnostic and therapeutic management of VTE is more challenging in the elderly. Therefore, we planned a randomized controlled trial on the efficacy of LMWH for the prevention of symptomatic VTE in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 70 years or older
* Admitted to hospital for an acute medical illness
* Anticipated duration of hospitalization of at least 4 days
* Life expectancy of at least 3 months

Exclusion Criteria:

* Admission for one of the following reasons:

  * Planned medical procedure.
  * Routine health assessment requiring admission for baseline/trending of health status (e.g., routine colonoscopy).
  * Admission encountered for another life circumstance that causes no bearing on health status and requires no medical intervention (e.g., lack of housing, economic inadequacy, care-giver respite, family circumstances, administrative).
* Hypersensitivity to heparin
* History of Heparin Induced Thrombocytopenia
* Active bleeding
* Bacterial endocarditis
* Platelet count of less than 80,000 per cubic millimeter
* Patients who require anticoagulant therapy for any indication, and those who received any type of anticoagulant therapy for > 48 hours
* Organic lesion prone to bleeding.
* Hemorrhagic events or bleeding tendency due to hemostasis disorders.
* Concomitant use of aspirin (> 160 mg/day), clopidogrel (> 75 mg/day), or of combined antiplatelet therapy
* Creatinine clearance < 15 ml/min
* Unable or unwilling to consent
* Ischemic stroke + hemorrhagic transformation
* Patient requiring admission to Intensive Care Unit

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2560 (Actual)
Dates: Start 2015-09-03 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
Occurence of the following events: symptomatic confirmed deep venous thrombosis (DVT), symptomatic confirmed pulmonary embolism (PE), or fatal PE | Occurence of any of the events through the Day 30 visit

SECONDARY OUTCOMES:
Occurence of the following events: Major bleeding, clinically relevant non major bleeding, symptomatic confirmed VTE (DVT or PE) or fatal PE, atherothrombotic cardiovascular events, cardiovascular death, Death from any cause. | Occurence of any of the events through the Day 30 and Day 90 visit
  The secondary outcomes is the occurrence of any of the following events:
  * Major bleeding as defined by the criteria of the International Society of Thrombosis and Haemostasis at day 30 and day 90
  * Clinically relevant non major bleeding and any bleeding at day 30 and day 90
  * Symptomatic confirmed VTE (DVT or PE) or fatal PE through the day 90 visit
  * Atherothrombotic cardiovascular events at day 30 and day 90
  * Cardiovascular death at day 30 and day 90
  * Death from any cause at day 30 and day 90
  * Rate of VTE and bleeding events at day 30 and day 90 according to creatinin clearance (< 50 ml/min and ≥ 50 ml/min), age range, D-dimer level and the use or not of antiplatelet therapy to identified the population at risk for VTE and bleeding.

CONTACTS AND LOCATIONS:
Locations (46):
- France (45):
  - Centre Hospitalier d'Agen, Agen
  - CHU Angers, Angers
  - CH Angoulême, Angoulême
  - CH d'Arras, Arras
  - CH Béthune, Béthune
  - Hôpital Jean Verdier (APHP), Bondy
  - CHU Bordeaux, Bordeaux
  - HIA Clermont-Tonnerre, Brest
  - CHRU Brest, Brest
  - CH Public du Cotentin, Cherbourg
  - CH Louis Mourier de Colombes, Colombes
  - CHU de Dijon, Dijon
  - CHU Grenoble, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - Groupe Hospitalier Le Havre, Le Havre
  - CHU Rouen, Le Petit-Quevilly
  - CHRU de Lille, Lille
  - CHU Limoges, Limoges
  - CHD Vendée - Site de Luçon, Luçon
  - Hôpital Edouard Herriot - CHU Lyon, Lyon
  - CHU Lyon, Lyon
  - Hôpital de la Timone - AP-HM, Marseille
  - Clinique Mutualiste Médico-chirurgical "Beau Soleil", Montpellier
  - CH des Pays de Morlaix, Morlaix
  - CHU Nancy, Nancy
  - CHU de Nantes, Nantes
  - Hôpital Cimiez - CHU Nice, Nice
  - HEGP - Paris, Paris
  - Hôpital Lariboisiere, Paris
  - Hôpital Saint-Antoine (APHP), Paris
  - Hôpital Broca- APHP, Paris
  - Hôpita Cochin - APHP, Paris
  - Institut Mutualiste Montsouris, Paris
  - CH Périgueux, Périgueux
  - CHU Poitiers, Poitiers
  - CH de Cornouaille - Quimper, Quimper
  - CHU Rennes, Rennes
  - Hôpital Charles Nicolle- CHU Rouen, Rouen
  - CHU La Réunion - Site Félix Guyon, Saint-Denis
  - CHU de Saint Etienne, Saint-Etienne
  - CHU La Réunion - site du GHSR, Saint-Pierre
  - CHRU Strasbourg- Service HTA et Maladies Vasculaires, Strasbourg
  - CHU Strasbourg - Service de Médecine Interne, Strasbourg
  - CH Intercommunal Toulon La Seyne sur Mer, Toulon
  - HIA Sainte-Anne Toulon, Toulon
- Hôpitaux Universitaires de Genève, Geneva, Switzerland

REFERENCES:
- [Derived] Mottier D, Girard P, Couturaud F, Lacut K, Le Moigne E, Paleiron N, Guellec D, Sanchez O, Cogulet V, Laporte S, Marhic G, Mismetti P, Presles E, Robert-Ebadi H, Mahe I, Plaisance L, Reny JL, Darbellay Farhoumand P, Cuvelier C, Le Henaff C, Lambert Y, Danguy des Deserts M, Rousseau Legrand C, Boutreux S, Bleher Y, Decours R, Trinh-Duc A, Armengol G, Benhamou Y, Daumas A, Guyot SL, De Carvalho H, Lamia B, Righini M, Meyer G, Le Gal G. Enoxaparin versus Placebo to Prevent Symptomatic Venous Thromboembolism in Hospitalized Older Adult Medical Patients. NEJM Evid. 2023 Aug;2(8):EVIDoa2200332. doi: 10.1056/EVIDoa2200332. Epub 2023 Jun 27. PMID 38320142